CLINICAL TRIAL: NCT03470818
Title: Applying Flipped Classroom Concepts to Simulation: the Effect of Pre-teaching Medical Content on Resident Acquisition and Retention of Non-technical Skills
Brief Title: Applying Flipped Learning Concepts to Simulation: the Effect on the Retention of Non-technical Skills
Acronym: FlippedSim
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 16.081
Record Dates: First submitted 2018-03-07; First posted 2018-03-20 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Crisis Resource Management; Flipped Classroom
Keywords: Medical Education; Flipped Classroom; Anxiety; Simulation; Achievement Emotions
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Preparatory instructional videos (flipped classroom model)
  32 participants
  Application of a flipped classroom model
  Prior to the simulation session, the intervention group will have received the study intervention. This consists in the provision of preparatory instruction about the medical knowledge required to complete the task work of the upcoming simulated acute care clinical situation. The format used to convey this off-loaded educational content will be short (approximately 15 minutes) narrated video PowerPoint presentations; every relevant medical situation incorporated in the simulation case will have a dedicated video presentation.
  These videos will be available to the intervention group participants on a web-based platform one week prior to the simulation session
  Interventions: Other: Preparatory instructional videos (flipped classroom model)
- Control group (Sham Comparator): Sham videos
  Participants in the control group will also be called to watch an online video prior to the simulation activity. However, this video presentation will not have any form of information regarding the upcoming simulation case; it will be an introductory video discussing the capacities of the simulation facility.
  This will limit any unwanted "snowball" effect where discussion between research participants could lead the control group participants to inquire about a video presentation that they would not exposed to.
  Interventions: Other: Sham video

INTERVENTIONS:
Other: Preparatory instructional videos (flipped classroom model) — The intervention consists in the provision of preparatory instruction about the medical knowledge required to complete the task work of the upcoming simulated acute care clinical situation. The format used to convey this off-loaded educational content will be short (approximately 15 minutes) narrated video PowerPoint presentations; every relevant medical situation incorporated in the simulation case will have a dedicated video presentation.
  These videos will be available to the intervention group participants on a web-based platform one week prior to the simulation session
  Arms: Intervention group
Other: Sham video — Participants in the control group will be called to watch an online video prior to the simulation activity. However, this video presentation will not have any form of information regarding the upcoming simulation case; it will be an introductory video discussing the capacities of the simulation facility. This will limit any unwanted "snowball" effect where discussion between research participants could lead the control group participants to inquire about a video presentation that they would not exposed to.
  Arms: Control group

SUMMARY:
The primary objective of this study is to assess if letting learners know in advance what medical illnesses will be practiced in an upcoming simulation session and providing them with instruction regarding that medical content ahead of time (flipped classroom model) will allow them to focus on the application of Crisis Resource Management (CRM) principles during a simulation session and result in an increase retention of theses skills. Secondary objectives of this study are to assess the relationship between the study intervention and learners' emotional responses and its impact on the retention of non-technical skills, in occurrence CRM

DETAILED DESCRIPTION:
The term "flipped classroom" refers to courses where basic educational content has been removed from the in-class schedule and has instead been provided in advance for learners to review prior to face-to-face interaction with the instructor. Consequently, during class time, learners use time ordinarily spent in lecture to instead practice applying their knowledge.

Although this methodology has been mainly described in classroom-based instruction, the underlying theory can conceptually apply to simulation training in the context of medical education. Too often, and especially with junior learners, time during simulation instruction is spent giving feedback directed at performance gaps caused by a lack of medical knowledge (e.g. medication dose, treatment plan, etc.). Unfortunately, teaching medical knowledge during debriefings takes away from the time spent practicing and discussing non-technical skills (NTS) such as communication, leadership, etc. If the objectives of a simulation session are directed towards increasing competencies in NTS (e.g., Crisis Resource Management [CRM]), efforts should be made to maximize the time spent on the application of these skills. Ensuring that learners possess the medical knowledge required to accomplish the task work of a case (e.g. diagnosis, treatment, etc.) beforehand could help focus their attention on teamwork competencies and result in educational gains.

The benefit of applying a flipped classroom model to simulation-based CRM instruction is anchored in two hypotheses:

1. The Cognitive Load Theory Hypothesis: Applying a flipped classroom model to CRM training could decrease the load imposed on learners' cognitive processes. According to this theory, working memory has a finite capacity and can only take on a certain load. When it is overloaded, new information cannot be processed and learning is impeded. Temporally separating the instructional content could help learners concentrate on the intended learning objectives of a simulation exercise designed to practice CRM skills. This could lead to enhanced proficiency and retention of these skills.
2. The Control Value Theory of Achievement Emotions Hypothesis: Achievement emotions are defined as emotions induced by learning activities or their outcomes. They are generated when performances of students are appraised according to a standard of excellence. Central to this theory is that "[…] individuals experience specific achievement emotions when they feel in control of, or out of control of, achievement activities and outcomes that are subjectively important to them […]". Negative emotions, such as anxiety, have been shown to reduce the cognitive resources available for learning. Providing preparatory instruction could regulate learners' stress response and reduce its impact on learning. In fact, increasing learners' knowledge of what will happen during simulation training can enhance their perceived control over the learning experience and limit the emergence of anticipatory anxiety. The act of sharing information prior to simulation training may also been seen as a gesture of transparency on the instructor's behalf. This has the potential to realign the perceived role of the instructor to a coaching instead of a judging role. A shared understanding of the upcoming learning experience may lessen socioevaluative anxiety by emphasizing the formative nature of the activity.

This study specifically tries to provide an answer to this research question: "Does providing preparatory instruction regarding the medical content of a simulation case to junior medical residents allow learners to focus more on Crisis Resource Management (CRM) principles thus resulting in an increase retention of Crisis Resource Management (CRM) skills three months after a technology-enhanced simulation session aimed at the acquisition of CRM competencies?"

The research question and underlying hypotheses will be tested in a between-subjects experimental design using a mixed-method approach. Subjects will be randomly allocated to an intervention (i.e. "flipped simulation") or a control group.

ELIGIBILITY:
Inclusion Criteria:

* First year residents in any surgical or medical specialty (including family medicine) that are required to achieve competencies in CRM skills per residency program requirements

Exclusion Criteria:

* endocrine disorders affecting cortisol metabolism (i.e., hypo/hyperthyroidism, Cushing's syndrome/disease, adrenal insufficiency, etc.)
* Corticosteroid therapy (except for topical)
* Use of drugs interfering with physiologic stress response (i.e., antidepressant medication, benzodiazepines, beta-blockers, calcium channel blockers, etc.)
* Pregnancy
* Knowledge of the simulation scenarios before study inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2018-01-19 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Overall Crisis Resource Management skills | Three months
  The between group difference in Crisis Resource Management skills three months post instruction measured by the overall Ottawa Crisis Resource Management Global Rating Scale mean score
  Scale ranges: 1 - 7
  Higher scores are associated with better performance

SECONDARY OUTCOMES:
Specific Crisis Resource Management skills | 3 months
  Difference in mean scores on the Ottawa Crisis Resource Management Global Rating Scale subcategories for the instructional and assessment sessions
  Scale ranges: 1 - 7
  Higher scores are associated with better performance
Stress response with salivary cortisol | Baseline and 3 months
  Between group difference in stress response (i.e. Peak minus baseline State Trait Anxiety Inventory score) during the instructional session and the learning assessment at 3 months
Stress response with State Trait Inventory Index | Baseline and 3 months
  Between group difference in stress response (i.e. Peak minus baseline State Trait Anxiety Inventory score) during the instructional session and the learning assessment at 3 months
Stress response difference with State Trait Anxiety Inventory | 3 months
  Between group difference in the mean change in stress response between the instructional session and the learning assessment at 3 months as measured by the State Trait Anxiety Inventory (i.e. State Trait Anxiety Inventory stress response for the assessment session minus the State Trait Anxiety Inventory stress response for the instructional session)
Stress response difference with salivary cortisol | 3 months
  Between group difference in the mean change in stress response between the instructional session and the learning assessment at 3 months as measured by cortisol levels (i.e. Cortisol stress response for the assessment session minus the cortisol stress response for the instructional session)
Emotional response assessed with the Achievement Emotion Questionnaire | Baseline and 3 months
  Between group difference in the incidence of specific achievement emotions before, during and after the Crisis Resource Management simulation training and the learning assessment at 3 months as specified in the Achievement Emotion Questionnaire
Qualitative assessment | Baseline and 3 months
  Differences in the qualitative themes obtained through semi-structure interviews for each groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No